CLINICAL TRIAL: NCT00141661
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase IIa, Multiple Dose, Multicenter Study in Subjects With Mild to Moderate Dementia of the Alzheimer's Type to Evaluate the Safety and Tolerability of Two 10-Week Dose Regimens of Orally-Administered PF-04494700
Brief Title: A Safety and Tolerability Evaluation of Two 10-Week Dose Regimens of Orally-Administered PF-04494700 in Alzheimer's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Trans Tech Pharmaceuticals (Unknown)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0341008; TTP488-201
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer Disease
Keywords: Interventional, Alzheimer, Safety and Tolerability
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose Arm (Experimental)
  Interventions: Drug: PF-04494700 - Low Dose Arm
- High Dose Arm (Experimental)
  Interventions: Drug: PF-04494700 - High Dose Arm
- Placebo Control (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: PF-04494700 - Low Dose Arm — 30 mg loading dose for 6 days, followed by 10 mg daily
  Arms: Low Dose Arm
Drug: PF-04494700 - High Dose Arm — 60 mg loading dose for 6 days, followed by 20 mg daily
  Arms: High Dose Arm
Drug: Placebo Comparator — Matching placebo.
  Arms: Placebo Control

SUMMARY:
A 10-week safety and tolerability study of a potential treatment for mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probably Alzheimer's disease for at least 1 year.
* Mini Mental State Exam (MMSE) score between 12-26 at screening.
* Participants must be receiving a cholinesterase inhibitor and/or memantine for at least 4 months, and on a stable dose for at least 2 months.

Exclusion Criteria:

* Current evidence of a neurological or psychiatric illness that could contribute to dementia.
* Living alone.
* Poorly controlled high blood pressure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety Measures include Adverse Events | Every Visit
Laboratory Tests | Every Office Visit
12-Lead Electrocardiogram | Every Office Visit
24-Hour 12-Lead Serial ECGs | Baseline, Study End

SECONDARY OUTCOMES:
Surrogate Efficacy Markers in Plasma: A-Beta, C-Reactive Protein, IL-1, IL-6, Isoprostanes, TNF-alpha, TNF-beta | Baseline, Visit 5, Study End
Cognitive Function Tests: ADAS-Cog, CDR-Sum of Boxes, MMSE, ADCS-ADL | Screening Visit, Baseline, Study End
Pharmacokinetic Profile | Baseline and Every Office Visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Memphis, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=TTP488-201&StudyName=A%20Safety%20and%20Tolerability%20%20Evaluation%20of%20Two%2010-Week%20Dose%20Regimens%20of%20Orally-Administereed%20PF-04494700%20in%20Alzheimer%27s%20Patients